# **School of Nursing**

# **LKS Faculty of Medicine**

# The University of Hong Kong

## Title:

The effects of the Buddy-Up Dyadic Physical Activity (BUDPA) Program on the health outcomes of care dyads of dementia: A pilot feasibility study

**Last Update: 1 November 2020** 

### School of Nursing, Li Ka Shing Faculty of Medicine, The University of Hong Kong

## **Information sheet (English version)**

#### **Study Title**

The effects of the Buddy-Up Dyadic Physical Activity (BUDPA) Program on the health outcomes of care dyads of dementia: A pilot feasibility study

#### Purpose of the study

The aim of this pilot study is to examine the feasibility and preliminary effect of a partnering exercise program on the health outcomes of the Patient with dementia and their family caregivers.

#### **Procedure**

You will be randomly assigned to receive either a partnering exercise program or usual care. Before you are assigned to either of these Program, the research assistant will use standardized questionnaires to assess cognitive function, neuro-psychiatric symptoms, and functional status of older adults with mild to early moderate dementia. For family caregivers of Patient with dementia, the research assistant will assess your caregiving burden, mood status and Positive Aspects of Caregiving.

For participants who join the partnering exercise program, a 12 weekly 1-hour training class is included. Each session starts with a 10-minute warm-up period using stretching exercise and stationary mobilizing exercise for trunk and limb joints at both upper and lower bodies (e.g. shoulders, elbows, wrists, hips, knees and ankles), and followed by a session of four to six selected partnering exercise, with duration increase gradually from 20 minutes to 40 minutes in four weeks in time. The Borg Rate of Perceived Exertion (Borg RPE) will be used to monitor the exercise intensity. The RA will explain the Borg RPE scale to you and instruct you to speed up or slow down your movements in order to achieve a feeling of 'somewhat hard' at the Borg RPE rating of 12-14. The training session will end with a 10-minute cool down session with walking exercise and stationary trunk and limb mobilizing exercise involving joints of shoulders, elbows, wrists, hips, knees, and ankles.

The first four weeks of training is mainly for conditioning and to develop the skills of the care dyads indoing the ten form of partnering exercise. From the fifth session onward, the care dyads are required to conduct the exercise self-practice for two more time at home. The RA will work out a goal attainment form for each care dyad, on which there is an exercise wheel to document the warm up, four self-selected forms of partnering exercise and the cool down to guide their self-practice. Relevant equipment such as elastic band and balls will be provided. In each subsequent week, the RA will invite your concerns about having the self-practice and to provide support accordingly. The goal attainment form will be revisited in the 8th and 12th week during the in-class exercise, and the care dyads are encouraged to re-select the exercise combination accordingly. A log-book will be provided to the care dyads to document the self- practice at home.

If you are assigned to join the Usual Care, activities will be provided by the elderly

community center such as dementia or caregiver supporting service.

No matter which type of program you are assigned to, another research assistant will give you telephone calls for 3 times (i.e., 6th, 12th and 18th week) to access your assess the health outcomes. The information will be used to conclude the effects of the Program you have received.

#### Risk and Benefits

The study intervention will not cause any pain, discomfort or harm to you. The exercise in the 12-week BUDPA Program is designed in accordance with the recommendations of the American College of Sports Medicine (ACSM)'s position stand on Exercise and Physical Activity for Older Adults. The training will follow the ACSM safety guidelines with assessment done on Blood Pressure, heart rate and contradictory symptoms prior to training. The major potential benefit is to improve cognitive outcomes of persons with dementia and manage the stress-related symptoms of their family caregivers

#### Anonymity, confidentially and nature of participation

All the collected data will be subject to strict anonymity and confidentiality. Your name will not appear on any data record sheets. They will be locked up in a secure location and only the researcher can have access. All the data will also be destroyed after use. Your participation is voluntary. You may refuse to participate or may withdraw consent and discontinue the participation in the study at any time. Your decision will not affect the quality of present or future care you receive in the hospital.

#### **Inquiry**

This study is undertaken by Prof. Doris YU. For any inquiry, please feel free to contact Prof. YU at 39176319.

You are cordially invited to participate in this study.

## School of Nursing, Li Ka Shing Faculty of Medicine, The University of Hong Kong

#### Informed consent

### Study Title:

The effects of the Buddy-Up Dyadic Physical Activity (BUDPA) Program on the health outcomes of care dyads of dementia: A pilot feasibility study

I hereby agree to participate in the above studies. I understand that the information obtained in the study will be used for future research and maybe published in academic literature.

I also know that if I disagree with the information obtained in the public study, I can continue to participate in the study. However, all personal data is kept strictly confidential and will not be made public. I understand all the benefits and risks associated with this study.

The researcher has explained the study to me in detail and asked me to ask questions and get a satisfactory reply. If I am involved in this study and cause any physical discomfort or emotional fluctuations, the researcher will treator refer to my treatment. I will not waive any legal rights by signing this consent form.

Ihereby signthis consent form to prove that all the information provided by me is correct. I understand that participation in this study is voluntary and I may withdraw this consent at any time without any reason, without affecting my current and future treatment.

I understand that my identity will be treated confidentially. I also allow the Institutional Review Board of the University of Hong Kong / Hospital Authority Hong Kong West Cluster and the relevant statutory bodies to directly check my research data to verify the relevant clinical research data, subject to the appropriate regulations and legislation and without infringing my privacy.

| Participant (PWD) signature | Participant (PWD) name | Date |
|-----------------------------------|-------------------------|------|
| Participant (Caregiver) signature | Proxy (Caregiver) name | Date |
| Research assistant signature | Research assistant name | Date |

After signing, I will receive a copy of the participating academic research materials page and signed informed consent for reservation.